CLINICAL TRIAL: NCT01305031
Title: Resuscitation of Late-preterm Infants by Using Room Air or 100% Oxygen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Director, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMU-FY2011-225, YKK10038
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Asphyxia
Keywords: Asphyxia; Resuscitation; Room Air
MeSH Terms: conditions — Asphyxia | interventions — Resuscitation; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Room air (Experimental): Initiation of resuscitation with 21% Oxygen, adjustments to the inspired oxygen concentration (increased 10%) will be made every 60 seconds for infants to achieve a target SpO2 range of 85-92%
  Interventions: Other: Resuscitation
- 100% Oxygen (Active Comparator): Initiation of resuscitation with 100% Oxygen and achieve oxygen saturation in the preset limits 85-92%
  Interventions: Other: 100% oxygen

INTERVENTIONS:
Other: Resuscitation — Use of inspiratory fraction of oxygen needed to achieve oxygen saturation in the preset limits 85-92%
  Arms: Room air
Other: 100% oxygen — Use of 100% oxygen needed to achieve oxygen saturation in the preset limits 85-92%
  Arms: 100% Oxygen

SUMMARY:
In this randomized control trial, the investigators hypothesize that late-preterm infants resuscitated with a "low oxygen delivery" strategy (initiation of resuscitation with room air) will result in a significant reduction in oxidant stress without any harmful clinical effects.

DETAILED DESCRIPTION:
The delivery of high oxygen concentrations leads to the production of free radicals that can injure many organ systems. Some studies have shown that resuscitation of term newborn infants with room air were safe and of great benefit. A static room air, however, may be inappropriate for resuscitation of preterm infants. The number of late-preterm infants has increased in recent years, which represent approximately 70% of all preterm infants. Our study will evaluate the safety and efficacy of using room air during resuscitation of late-preterm infants and whether this will avoid oxidative stress derived damage and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* inborn infant
* gestation 34 weeks to 36 weeks 6 days

Exclusion Criteria:

• known chromosomal or congenital anomalies

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
oxidative stress status | 7 days
oxygen saturations | 10 min

SECONDARY OUTCOMES:
Days on oxygen | 28 days
Days on conventional ventilation | 28 days
Days on high frequency ventilation | 28 days
Days on nasal canula | 28 days
Pneumothorax | 28 days
Oxygen requirement | At 36 weeks adjusted age
Patent ductus arteriosus | 28 days
Necrotizing Enterocolitis | 28 days
Intracranial hemorrhage | 28 days
Hypoxic ischemic encephalopathy | 28 days
Retinopathy of prematurity | 28 days
Death | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Shuping Han, PhD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China